CLINICAL TRIAL: NCT00366678
Title: A Phase 3, Randomized, Active-Controlled, Double-blind Trial Evaluating the Safety, Tolerability, and Immunogenicity of a 13-valent Pneumococcal Conjugate Vaccine in Healthy Infants Given With Routine Pediatric Vaccinations in France.
Brief Title: Study to Evaluate a 13-valent Pneumococcal Conjugate Vaccine in Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6096A1-008
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Results first posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-07

CONDITIONS: Vaccines, Pneumococcal
Keywords: Safety; Vaccine
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine; Pentavac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 13-valent pneumococcal conjugate vaccine (Experimental): 13-valent pneumococcal conjugate vaccine
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine; Drug: Pentavac
- 7-valent pneumococcal conjugate vaccine (Active Comparator): 7-valent pneumococcal conjugate vaccine
  Interventions: Biological: 7-valent pneumococcal conjugate vaccine; Drug: Pentavac

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — Single 0.5 mL dose given at 2, 3, 4, and 12 months of age.
  Arms: 13-valent pneumococcal conjugate vaccine
Biological: 7-valent pneumococcal conjugate vaccine — Single 0.5 mL dose given at 2, 3, 4, and 12 months of age.
  Arms: 7-valent pneumococcal conjugate vaccine
Drug: Pentavac — The Pentavac was administered by intramuscular injection 0.5 ml into the anterolateral thigh muscle of the right leg at 2, 3, and 4 months (infant series) and 12 months of age (toddler dose).

SUMMARY:
The purpose of this study is to assess the safety, tolerability and immunogenicity of a 13-valent pneumococcal conjugate (13vPnC) vaccine compared to Prevenar (7vPnC), when given concomitantly with routine pediatric vaccines in France.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 2-month-old infants.
* Available for the entire study period.

Exclusion criteria:

· Known contraindication to vaccines.

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 613 (Actual)
Dates: Start 2006-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For France, infomedfrance@wyeth.com
Locations (43):
- France (43):
  - Albi
  - Amiens
  - Ancenis
  - Blanquefort
  - Bondues
  - Bordeaux
  - Brest
  - Châlons-en-Champagne
  - Créteil
  - Dijon
  - Draguignan
  - Essey-lès-Nancy
  - Écully
  - Floirac
  - Fréjus
  - Garges-lès-Gonesse
  - Illkirch-Graffenstaden
  - Joué-lès-Tours
  - Le Havre
  - Le Plessis-Trévise
  - Le Pontet
  - Les Lilas
  - Les Sables-d'Olonne
  - Libourne
  - Lingolsheim
  - Lyon
  - Marcq-en-Barœul
  - Maromme
  - Moûtiers
  - Nancy
  - Nice
  - Nogent-sur-Marne
  - Oullins
  - Paris
  - Rouen
  - Strasbourg
  - Thionville
  - Tours
  - Tresses Melac
  - Vandœuvre-lès-Nancy
  - Vaulx-en-Velin
  - Villeneuve-d'Ascq
  - Vitry-sur-Seine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in France from October 2006 to July 2007.
Pre-assignment Details: Participants were enrolled into the study according to inclusion/exclusion criteria without a screening period.
Groups:
- 13vPnC/13vPnC Vaccine: Participants received one single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with a vaccine containing diphtheria, tetanus, 2-component pertussis (DTaP), inactivated poliovirus (IPV), and hemophilus influenza type b vaccines (Hib) (Pentavac) at 2, 3, and 4 months of age (infant series) and 12 months of age (toddler dose).
- 7vPnC/7vPnC Vaccine: Participants received one single 0.5 milliliter (mL) dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with a vaccine containing diphtheria, tetanus, 2-component pertussis (DTaP), inactivated poliovirus (IPV), and hemophilus influenza type b vaccines (Hib) (Pentavac) at 2, 3, and 4 months of age (infant series) and 12 months of age (toddler dose).
- 7vPnC/13vPnC Vaccine: Participants received one single 0.5 milliliter (mL) dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with a vaccine containing diphtheria, tetanus, 2-component pertussis (DTaP), inactivated poliovirus (IPV), and hemophilus influenza type b vaccines (Hib) (Pentavac) at 2, 3, and 4 months of age (infant series). Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC)coadministered with Pentavac at 12 months of age (toddler dose).
Period: Infant Series
Arm/Group | 13vPnC/13vPnC Vaccine | 7vPnC/7vPnC Vaccine | 7vPnC/13vPnC Vaccine
Started | 304 | 309 | 0
Vaccinated Dose 1 | 302 | 309 | 0
Vaccinated Dose 2 | 295 | 304 | 0
Vaccinated Dose 3 | 291 | 302 | 0
Completed | 290 | 299 | 0
Not Completed | 14 | 10 | 0
Not completed — Withdrawal by Subject | 8 | 6 | 0
Not completed — Protocol Violation | 4 | 3 | 0
Not completed — Failed to return | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: After Infant
Arm/Group | 13vPnC/13vPnC Vaccine | 7vPnC/7vPnC Vaccine | 7vPnC/13vPnC Vaccine
Started | 290 | 299 | 0
Completed | 273 | 289 | 0
Not Completed | 17 | 10 | 0
Not completed — Withdrawal by Subject | 8 | 4 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Failed to return | 5 | 5 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Period: Toddler Dose
Arm/Group | 13vPnC/13vPnC Vaccine | 7vPnC/7vPnC Vaccine | 7vPnC/13vPnC Vaccine
Started | 273 | 152 | 137
Completed | 268 | 151 | 137
Not Completed | 5 | 1 | 0
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Failed to return | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — protocol deviation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC/13vPnC Vaccine | 7vPnC/7vPnC Vaccine | Total
Number analyzed (Participants) | 304 | 309 | 613
Age Continuous [Mean (Standard Deviation); unit: months] | 2.1 (0.5) | 2.1 (0.5) | 2.1 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 164 | 333
  Male | 135 | 145 | 280

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Predefined Antibody Levels for Diphtheria, Tetanus, Hemophilus Influenza Type b (Hib), Poliomyelitis (Type 1, 2, 3), Pertussis Toxin (PT) and Filamentous Hemagglutinin (FHA) in 13vPnC Group Relative to 7vPnC Group
Description: Percentage of participants achieving predefined antibody threshold levels ≥0.1 IU/mL for diphtheria, ≥0.1 IU/mL for tetanus, ≥ 0.15 μg/mL for Hib polyribosylribitol phosphate (PRP), antibody titer ≥1:8 for polio and ≥5 EU/mL for pertussis (PT and FHA) with the corresponding 95% CI for each concomitant antigen are presented.
Time Frame: One Month After the 3-Dose Infant Series (at 5 months of age) and the Toddler Dose (at 13 months of age)
Population: The evaluable immunogenicity (per protocol) population was the primary analysis population consisting of eligible subjects who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC After the Infant Series; 13vPnC After the Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with a vaccine containing Pentavac at 2, 3, and 4 months of age (infant series) and 12 months of age (toddler dose).
- 7vPnC After the Infant Series; 7vPnC After the Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with a vaccine containing Pentavac at 2, 3, and 4 months of age (infant series) and 12 months of age (toddler dose).
Arm/Group | 13vPnC After the Infant Series | 7vPnC After the Infant Series | 13vPnC After the Toddler Dose | 7vPnC After the Toddler Dose
Number analyzed (Participants) | 266 | 263 | 241 | 133
percentage of participants
  Pertussis - PT Infant ≥5 Toddler 5 (EU/mL) | 100.0 [98.6 to 100.0] | 100.0 [98.6 to 100.0] | 100.0 [98.5 to 100.0] | 100.0 [97.3 to 100.0]
  Pertussis - PT Infant ≥26 Toddler 17 (EU/mL) | 94.3 [90.8 to 96.8] | 95.0 [91.7 to 97.3] | 98.3 [95.8 to 99.5] | 96.2 [91.4 to 98.8]
  Pertussis - FHA Infant ≥5 Toddler 5 (EU/mL) | 100.0 [98.6 to 100.0] | 100.0 [98.6 to 100.0] | 100.0 [98.5 to 100.0] | 100.0 [97.3 to 100.0]
  Pertussis - FHA Infant ≥7.82 Toddler 7.82 (EU/mL) | 100.0 [98.6 to 100.0] | 100.0 [98.6 to 100.0] | 100.0 [98.5 to 100.0] | 100.0 [97.3 to 100.0]
  Pertussis - FHA Infant ≥36.00 Toddler 75 (EU/mL) | 93.5 [89.9 to 96.2] | 95.8 [92.6 to 97.9] | 92.5 [88.4 to 95.5] | 95.5 [90.4 to 98.3]
  Diphtheria 0.1 (IU/mL) | 76.5 [70.9 to 81.5] | 84.6 [79.6 to 88.7] | 99.2 [97.0 to 99.9] | 100 [97.3 to 100.0]
  Diphtheria 0.01 (IU/mL) | 100.0 [98.6 to 100.0] | 100.0 [98.6 to 100.0] | 100.0 [98.5 to 100.0] | 100.0 [97.3 to 100.0]
  Tetanus 0.1 (IU/mL) | 84.9 [80.0 to 89.1] | 82.2 [76.9 to 86.7] | 96.2 [93.0 to 98.3] | 98.5 [94.7 to 99.8]
  Tetanus 0.01 (IU/mL) | 100.0 [98.6 to 100.0] | 100.0 [98.6 to 100.0] | 100.0 [98.5 to 100.0] | 100.0 [97.3 to 100.0]
  Polio Type 1 (1:8) | 88.8 [84.3 to 92.3] | 91.0 [86.8 to 94.2] | 97.9 [95.2 to 99.3] | 98.4 [94.5 to 99.8]
  Polio Type 2 (1:8) | 77.7 [72.1 to 82.6] | 82.0 [76.8 to 86.5] | 98.7 [96.4 to 99.7] | 99.2 [95.8 to 100.0]
  Polio Type 3 (1:8) | 92.6 [88.7 to 95.5] | 93.0 [89.1 to 95.8] | 99.2 [97.0 to 99.9] | 100.0 [97.2 to 100.0]
  Hib (PRP) 0.15 (μg/mL) | 95.5 [92.1 to 97.7] | 94.6 [91.0 to 97.1] | 100.0 [98.5 to 100.0] | 100.0 [97.2 to 100.0]
  Hib (PRP) 1.0 (μg/mL) | 58.6 [52.1 to 64.9] | 63.1 [56.6 to 69.2] | 97.9 [95.2 to 99.3] | 97.7 [93.5 to 99.5]
Statistical Analysis 1: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Pertussis - PT the difference in percentages between the two groups (13vPnC - 7vPnC) at (≥5 EU/mL) threshold was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lowest limit of 2-sided 95% CI for the difference between the 2 groups (13vPnC - 7vPnC) > -10%; Difference = 0.0, 95% CI [-1.4 to 1.4]
Statistical Analysis 2: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Pertussis - PTf the difference in percentages between the two groups (13vPnC - 7vPnC) at (≥26.00 EU/mL) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -0.7, 95% CI [-4.8 to 3.3]
Statistical Analysis 3: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Pertussis - FHA the difference in percentages between the two groups (13vPnC - 7vPnC) at (≥5 EU/mL) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-1.4 to 1.4]
Statistical Analysis 4: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Pertussis - FHAf the difference in percentages between the two groups (13vPnC - 7vPnC) at (≥36.00 EU/mL) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -2.3, 95% CI [-6.4 to 1.7]
Statistical Analysis 5: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Pertussis - FHA the difference in percentages between the two groups (13vPnC - 7vPnC) at (≥7.82 EU/mL) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-1.4 to 1.4]
Statistical Analysis 6: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Pertussis - PT the difference in percentages between the two groups (13vPnC - 7vPnC) at (5 EU/mL) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-1.7 to 2.7]
Statistical Analysis 7: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Pertussis - PTf the difference in percentages between the two groups (13vPnC - 7vPnC) at (17.00 EU/mL) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 2.1, 95% CI [-1.4 to 6.8]
Statistical Analysis 8: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Pertussis - FHA the difference in percentages between the two groups (13vPnC - 7vPnC) at (5 EU/mL) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-1.7 to 2.7]
Statistical Analysis 9: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Pertussis - FHA the difference in percentages between the two groups (13vPnC - 7vPnC) at (7.82 EU/mL) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-1.7 to 2.7]
Statistical Analysis 10: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Pertussis - FHAf the difference in percentages between the two groups (13vPnC - 7vPnC) at (75.00 EU/mL) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -3.0, 95% CI [-8.0 to 2.5]
Statistical Analysis 11: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Diphtheria the difference in percentages between the two groups (13vPnC - 7vPnC) at 0.1 (IU/mL) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -8.0, 95% CI [-14.9 to -1.2]
Statistical Analysis 12: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Diphtheria the difference in percentages between the two groups (13vPnC - 7vPnC) at 0.01 (IU/mL) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-1.4 to 1.4]
Statistical Analysis 13: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Tetanus the difference in percentages between the two groups (13vPnC - 7vPnC) at 0.1 (IU/mL) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 2.7, 95% CI [-3.7 to 9.2]
Statistical Analysis 14: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Tetanus the difference in percentages between the two groups (13vPnC - 7vPnC) at 0.01 (IU/mL) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-1.5 to 1.5]
Statistical Analysis 15: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; [analysis description as in outcome 1, analysis 11]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -0.8, 95% CI [-3.1 to 1.8]
Statistical Analysis 16: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; [analysis description as in outcome 1, analysis 12]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-1.7 to 2.7]
Statistical Analysis 17: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; [analysis description as in outcome 1, analysis 13]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -2.3, 95% CI [-5.8 to 1.8]
Statistical Analysis 18: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; [analysis description as in outcome 1, analysis 14]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-1.7 to 2.7]
Statistical Analysis 19: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Polio Type 1 the difference in percentages between the two groups (13vPnC - 7vPnC) at (1:8) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -2.3, 95% CI [-7.6 to 3.0]
Statistical Analysis 20: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Polio Type 2 the difference in percentages between the two groups (13vPnC - 7vPnC) at (1:8) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -4.3, 95% CI [-11.4 to 2.6]
Statistical Analysis 21: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Polio Type 3 the difference in percentages between the two groups (13vPnC - 7vPnC) at (1:8) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -0.3, 95% CI [-5.0 to 4.3]
Statistical Analysis 22: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; [analysis description as in outcome 1, analysis 19]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -0.5, 95% CI [-3.6 to 3.5]
Statistical Analysis 23: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; [analysis description as in outcome 1, analysis 20]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -0.5, 95% CI [-3.1 to 3.0]
Statistical Analysis 24: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; [analysis description as in outcome 1, analysis 21]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -0.8, 95% CI [-3.1 to 1.9]
Statistical Analysis 25: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Hib (PRP) the difference in percentages between the two groups (13vPnC - 7vPnC) at 0.15 (μg/mL) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.9, 95% CI [-3.2 to 5.0]
Statistical Analysis 26: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Hib (PRP) the difference in percentages between the two groups (13vPnC - 7vPnC) at 1.0 (μg/mL) threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -4.5, 95% CI [-13.2 to 4.4]
Statistical Analysis 27: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; [analysis description as in outcome 1, analysis 25]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-1.7 to 2.8]
Statistical Analysis 28: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; [analysis description as in outcome 1, analysis 26]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.2, 95% CI [-3.1 to 4.5]

2. Secondary Outcome: Percentage of Participants Achieving a Pneumococcal Antibody Level ≥0.35µg/mL (ELISA) After the Toddler Dose in the 13vPnC/13vPnC, 7vPnC/7vPnC and 7vPnC/13vPnC Groups
Description: Percentages of participants achieving World health Organization (WHO) predefined antibody threshold ≥0.35μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after the toddler dose (at 13 months of age)
Population: Evaluable immunogenicity (per protocol) population who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n) = number of participants with a determinate antibody concentration for the specified serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC Infant Series / 13vPnC Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with a vaccine containing Pentavac at 2, 3, and 4 months of age (infant series) and 12 months of age (toddler dose).
- 7vPnC Infant Series / 7vPnC Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with a vaccine containing Pentavac at 2, 3, and 4 months of age (infant series) and 12 months of age (toddler dose).
- 7vPnC Infant Series / 13vPnC Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with Pentavac at 2, 3, and 4 months. One single 0.5 mL dose of 13vPnC was coadministered with Pentavac at 12 months of age.
Arm/Group | 13vPnC Infant Series / 13vPnC Toddler Dose | 7vPnC Infant Series / 7vPnC Toddler Dose | 7vPnC Infant Series / 13vPnC Toddler Dose
Number analyzed (Participants) | 241 | 133 | 121
percentage of participants
  Common Serotypes - Serotype 4 (n=233,126,111) | 100.0 [98.4 to 100.0] | 100.0 [97.1 to 100.0] | 99.1 [95.1 to 100.0]
  Common Serotypes - Serotype 6B (n=233,126,108) | 99.6 [97.6 to 100.0] | 99.2 [95.7 to 100.0] | 98.1 [93.5 to 99.8]
  Common Serotypes - Serotype 9V (n=232,124,109) | 100.0 [98.4 to 100.0] | 100.0 [97.1 to 100.0] | 100.0 [96.7 to 100.0]
  Common Serotypes - Serotype 14 (n=233,135,111) | 99.6 [97.6 to 100.0] | 100.0 [97.1 to 100.0] | 99.1 [95.1 to 100.0]
  Common Serotypes - Serotype 18C (n=230,125,113) | 99.6 [97.6 to 100.0] | 99.2 [95.6 to 100.0] | 98.2 [93.8 to 99.8]
  Common Serotypes - Serotype 19F (n=233,126,112) | 97.9 [95.1 to 99.3] | 97.6 [93.2 to 99.5] | 97.3 [92.4 to 99.4]
  Common Serotypes - Serotype 23F (n=232,123,111) | 99.6 [97.6 to 100.0] | 99.2 [95.6 to 100.0] | 99.1 [95.1 to 100.0]
  Additional Serotypes - Serotype 1 (n=233,119,112) | 100.0 [98.4 to 100.0] | 0.8 [0.0 to 4.6] | 95.5 [89.9 to 98.5]
  Additional Serotypes - Serotype 3 (n=233,124,113) | 94.8 [91.2 to 97.3] | 13.7 [8.2 to 21.0] | 93.8 [87.7 to 97.5]
  Additional Serotypes - Serotype 5 (n=236,111,111) | 100.0 [98.4 to 100.0] | 73.0 [63.7 to 81.0] | 90.1 [83.0 to 94.9]
  Additional Serotypes - Serotype 6A (n=235,124,109) | 100.0 [98.4 to 100.0] | 89.5 [82.7 to 94.3] | 89.9 [82.7 to 94.9]
  Additional Serotypes - Serotype 7F (n=234,124,110) | 100.0 [98.4 to 100.0] | 7.3 [3.4 to 13.3] | 100.0 [96.7 to 100.0]
  Additional Serotypes - Serotype 19A(n=233,127,112) | 100.0 [98.4 to 100.0] | 100.0 [97.1 to 100.0] | 100.0 [96.8 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC Infant Series / 13vPnC Toddler Dose vs 7vPnC Infant Series / 7vPnC Toddler Dose; For serotype 4 the difference in percentages between the two groups (13vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 7vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = 0.0, 95% CI [-1.7 to 2.9]
Statistical Analysis 2: Comparison: 13vPnC Infant Series / 13vPnC Toddler Dose vs 7vPnC Infant Series / 13vPnC Toddler Dose; For serotype 4 the difference in percentages between the two groups (13vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 13vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = 0.9, 95% CI [-0.9 to 4.9]
Statistical Analysis 3: Comparison: 7vPnC Infant Series / 7vPnC Toddler Dose vs 7vPnC Infant Series / 13vPnC Toddler Dose; For serotype 4 the difference in percentages between the two groups (7vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 7vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = -0.9, 95% CI [-4.9 to 2.1]
Statistical Analysis 4: Comparison: 13vPnC Infant Series / 13vPnC Toddler Dose vs 7vPnC Infant Series / 7vPnC Toddler Dose; For serotype 6B the difference in percentages between the two groups (13vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 7vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = 0.4, 95% CI [-1.8 to 3.8]
Statistical Analysis 5: Comparison: 13vPnC Infant Series / 13vPnC Toddler Dose vs 7vPnC Infant Series / 13vPnC Toddler Dose; For serotype 6B the difference in percentages between the two groups (13vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 13vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = 1.4, 95% CI [-1.1 to 5.9]
Statistical Analysis 6: Comparison: 7vPnC Infant Series / 7vPnC Toddler Dose vs 7vPnC Infant Series / 13vPnC Toddler Dose; For serotype 6B the difference in percentages between the two groups (7vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 7vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = -1.1, 95% CI [-5.8 to 2.7]
Statistical Analysis 7: Comparison: 13vPnC Infant Series / 13vPnC Toddler Dose vs 7vPnC Infant Series / 7vPnC Toddler Dose; For serotype 9V the difference in percentages between the two groups (13vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 7vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = 0.0, 95% CI [-1.7 to 2.9]
Statistical Analysis 8: Comparison: 13vPnC Infant Series / 13vPnC Toddler Dose vs 7vPnC Infant Series / 13vPnC Toddler Dose; For serotype 9V the difference in percentages between the two groups (13vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 13vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = 0.0, 95% CI [-1.8 to 3.3]
Statistical Analysis 9: Comparison: 7vPnC Infant Series / 7vPnC Toddler Dose vs 7vPnC Infant Series / 13vPnC Toddler Dose; For serotype 9V the difference in percentages between the two groups (7vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 7vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = 0.0, 95% CI [-3.3 to 3.0]
Statistical Analysis 10: Comparison: 13vPnC Infant Series / 13vPnC Toddler Dose vs 7vPnC Infant Series / 7vPnC Toddler Dose; For serotype 14 the difference in percentages between the two groups (13vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 7vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = -0.4, 95% CI [-2.5 to 2.4]
Statistical Analysis 11: Comparison: 13vPnC Infant Series / 13vPnC Toddler Dose vs 7vPnC Infant Series / 13vPnC Toddler Dose; For serotype 14 the difference in percentages between the two groups (13vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 13vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = 0.5, 95% CI [-1.8 to 4.4]
Statistical Analysis 12: Comparison: 7vPnC Infant Series / 7vPnC Toddler Dose vs 7vPnC Infant Series / 13vPnC Toddler Dose; For serotype 14 the difference in percentages between the two groups (7vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 7vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = -0.9, 95% CI [-4.9 to 2.1]
Statistical Analysis 13: Comparison: 13vPnC Infant Series / 13vPnC Toddler Dose vs 7vPnC Infant Series / 7vPnC Toddler Dose; For serotype 18C the difference in percentages between the two groups (13vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 7vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = 0.4, 95% CI [-1.8 to 3.8]
Statistical Analysis 14: Comparison: 13vPnC Infant Series / 13vPnC Toddler Dose vs 7vPnC Infant Series / 13vPnC Toddler Dose; For serotype 18C the difference in percentages between the two groups (13vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 13vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = 1.3, 95% CI [-1.1 to 5.7]
Statistical Analysis 15: Comparison: 7vPnC Infant Series / 7vPnC Toddler Dose vs 7vPnC Infant Series / 13vPnC Toddler Dose; For serotype 18C the difference in percentages between the two groups (7vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 7vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = -1.0, 95% CI [-5.5 to 2.8]
Statistical Analysis 16: Comparison: 13vPnC Infant Series / 13vPnC Toddler Dose vs 7vPnC Infant Series / 7vPnC Toddler Dose; For serotype 19F the difference in percentages between the two groups (13vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 7vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = 0.2, 95% CI [-3.1 to 4.7]
Statistical Analysis 17: Comparison: 13vPnC Infant Series / 13vPnC Toddler Dose vs 7vPnC Infant Series / 13vPnC Toddler Dose; For serotype 19F the difference in percentages between the two groups (13vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 13vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = 0.5, 95% CI [-2.9 to 5.4]
Statistical Analysis 18: Comparison: 7vPnC Infant Series / 7vPnC Toddler Dose vs 7vPnC Infant Series / 13vPnC Toddler Dose; For serotype 19F the difference in percentages between the two groups (7vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 7vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = -0.3, 95% CI [-5.5 to 4.4]
Statistical Analysis 19: Comparison: 13vPnC Infant Series / 13vPnC Toddler Dose vs 7vPnC Infant Series / 7vPnC Toddler Dose; For serotype 23F the difference in percentages between the two groups (13vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 7vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = 0.4, 95% CI [-1.8 to 3.9]
Statistical Analysis 20: Comparison: 13vPnC Infant Series / 13vPnC Toddler Dose vs 7vPnC Infant Series / 13vPnC Toddler Dose; For serotype 23F the difference in percentages between the two groups (13vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 13vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = 0.5, 95% CI [-1.9 to 4.4]
Statistical Analysis 21: Comparison: 7vPnC Infant Series / 7vPnC Toddler Dose vs 7vPnC Infant Series / 13vPnC Toddler Dose; For serotype 23F the difference in percentages between the two groups (7vPnC Infant Series / 13vPnC Toddler Dose - 7vPnC Infant Series / 7vPnC Toddler Dose) was calculated; Test type: Superiority or Other; Difference = -0.1, 95% CI [-4.1 to 3.7]

3. Secondary Outcome: Pneumococcal Geometric Mean Concentration (GMC) Before and After the Toddler Dose in the 13vPnC/13vPnC, 7vPnC/7vPnC and 7vPnC/13vPnC Groups
Description: Antibody GMC as measured by ELISA for 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after the Toddler Dose (at 13 months of age)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Groups:
- 13vPnC/13vPnC Before Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with a vaccine containing Pentavac at 2, 3, and 4 months of age (infant series) and 12 months of age (toddler dose).
- 13vPnC/13vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with a vaccine containing Pentavac at 2, 3, and 4 months of age (infant series) and 12 months of age (toddler dose), assessment made at 13 months of age.
- 7vPnC/7vPnC Before Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with a vaccine containing Pentavac at 2, 3, and 4 months of age (infant series) and 12 months of age (toddler dose).
- 7vPnC/7vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with a vaccine containing Pentavac at 2, 3, and 4 months of age (infant series) and 12 months of age (toddler dose), assessment made at 13 months of age.
- 7vPnC/13vPnC Before Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with Pentavac at 2, 3, and 4 months of age (infant series). Participants recieved one single 0.5 mL dose of 13vPnC coadministered with Pentavac at 12 months of age (toddler dose).
- 7vPnC/13vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with Pentavac at 2, 3, and 4 months of age (infant series). Participants received one single 0.5 mL dose of 13vPnC coadministered with Pentavac at 12 months of age (toddler dose), assessment made at 13 months of age.
Arm/Group | 13vPnC/13vPnC Before Toddler Dose | 13vPnC/13vPnC After Toddler Dose | 7vPnC/7vPnC Before Toddler Dose | 7vPnC/7vPnC After Toddler Dose | 7vPnC/13vPnC Before Toddler Dose | 7vPnC/13vPnC After Toddler Dose
Number analyzed (Participants) | 241 | 241 | 133 | 133 | 121 | 121
μg/mL
  Common - Serotype 4 (n=239,233,131,126,118,111) | 0.3 [0.3 to 0.3] | 4.2 [3.8 to 4.7] | 0.5 [0.4 to 0.5] | 4.8 [4.2 to 5.6] | 0.5 [0.4 to 0.5] | 4.0 [3.4 to 4.8]
  Common - Serotype 6B (n=235,233,131,126,115,108) | 1.0 [0.9 to 1.1] | 9.0 [8.0 to 10.1] | 1.1 [0.9 to 1.3] | 9.6 [8.3 to 11.2] | 0.9 [0.8 to 1.1] | 10.3 [8.2 to 13.0]
  Common - Serotype 9V (n=239,232,131,124,118,109) | 0.4 [0.4 to 0.5] | 2.3 [2.3 to 2.8] | 0.5 [0.5 to 0.6] | 3.2 [2.8 to 3.7] | 0.4 [0.4 to 0.5] | 2.3 [2.0 to 2.6]
  Common - Serotype 14 (n=238,233,131,125,118,111) | 2.0 [1.8 to 2.3] | 9.5 [8.5 to 10.6] | 2.4 [2.1 to 2.9] | 10.8 [9.4 to 12.5] | 2.4 [2.0 to 3.0] | 7.8 [6.6 to 9.3]
  Common - Serotype 18C (n=239,230,131,125,118,113) | 0.3 [0.3 to 0.3] | 2.3 [2.1 to 2.5] | 0.3 [0.3 to 0.4] | 2.8 [2.5 to 3.2] | 0.3 [0.3 to 0.4] | 2.4 [2.0 to 2.9]
  Common - Serotype 19F (n=239,233,130,126,118,112) | 0.7 [0.6 to 0.7] | 5.2 [4.5 to 6.0] | 0.7 [0.6 to 0.9] | 4.1 [3.4 to 5.0] | 0.6 [0.5 to 0.7] | 3.7 [3.0 to 4.6]
  Common - Serotype 23F (n=237,232,130,123,118,111) | 0.3 [0.2 to 0.3] | 3.0 [2.7 to 3.4] | 0.3 [0.3 to 0.4] | 3.7 [3.1 to 4.3] | 0.3 [0.2 to 0.4] | 3.1 [2.6 to 3.7]
  Additional-Serotype 1 (n=239,233,128,119,116,112) | 0.4 [0.4 to 0.5] | 4.1 [3.7 to 4.5] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 1.8 [1.5 to 2.2]
  Additional-Serotype 3 (n=232,233,128,124,115,113) | 0.2 [0.2 to 0.2] | 1.0 [0.9 to 1.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 1.3 [1.1 to 1.5]
  Additional-Serotype 5 (n=236,236,128,124,115,113) | 0.8 [0.7 to 0.9] | 3.3 [3.0 to 3.7] | 0.4 [0.4 to 0.5] | 0.5 [0.4 to 0.6] | 0.4 [0.4 to 0.5] | 1.1 [1.0 to 1.3]
  Additional-Serotype 6A (n=238,235,122,124,116,109) | 0.9 [0.8 to 1.0] | 6.1 [5.5 to 6.8] | 0.4 [0.3 to 0.5] | 1.5 [1.3 to 1.9] | 0.4 [0.3 to 0.4] | 2.6 [2.0 to 3.4]
  Additional-Serotype 7F (n=239,234,131,124,117,110) | 0.8 [0.7 to 0.9] | 4.5 [4.1 to 5.0] | 0.1 [0.0 to 0.1] | 0.1 [0.0 to 0.1] | 0.1 [0.1 to 0.1] | 3.7 [3.2 to 4.3]
  Additional-Serotype 19A(n=237,233,131,127,117,112) | 1.5 [1.3 to 1.7] | 9.5 [8.5 to 10.6] | 1.1 [0.9 to 1.3] | 4.0 [3.5 to 4.5] | 0.9 [0.7 to 1.1] | 5.3 [4.6 to 6.2]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC After Toddler Dose vs 7vPnC/7vPnC After Toddler Dose; For serotype 4 after the toddler dose the GMC ratio (13vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/7vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 0.87, 95% CI [0.73 to 1.03]
Statistical Analysis 2: Comparison: 7vPnC/7vPnC After Toddler Dose vs 7vPnC/13vPnC After Toddler Dose; For serotype 4 after the toddler dose the GMC ratio (7vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/7vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 0.83, 95% CI [0.67 to 1.03]
Statistical Analysis 3: Comparison: 13vPnC/13vPnC After Toddler Dose vs 7vPnC/13vPnC After Toddler Dose; For serotype 4 after the toddler dose the GMC ratio (13vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 1.04, 95% CI [0.86 to 1.26]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC After Toddler Dose vs 7vPnC/7vPnC After Toddler Dose; For serotype 6B after the toddler dose the GMC ratio (13vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/7vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 0.93, 95% CI [0.77 to 1.13]
Statistical Analysis 5: Comparison: 7vPnC/7vPnC After Toddler Dose vs 7vPnC/13vPnC After Toddler Dose; For serotype 6B after the toddler dose the GMC ratio (7vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/7vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 1.07, 95% CI [0.82 to 1.40]
Statistical Analysis 6: Comparison: 13vPnC/13vPnC After Toddler Dose vs 7vPnC/13vPnC After Toddler Dose; For serotype 6B after the toddler dose the GMC ratio (13vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 0.87, 95% CI [0.69 to 1.10]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC After Toddler Dose vs 7vPnC/7vPnC After Toddler Dose; For serotype 9V after the toddler dose the GMC ratio (13vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/7vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 0.80, 95% CI [0.68 to 0.94]
Statistical Analysis 8: Comparison: 7vPnC/7vPnC After Toddler Dose vs 7vPnC/13vPnC After Toddler Dose; For serotype 9V after the toddler dose the GMC ratio (7vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/7vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 0.71, 95% CI [0.59 to 0.85]
Statistical Analysis 9: Comparison: 13vPnC/13vPnC After Toddler Dose vs 7vPnC/13vPnC After Toddler Dose; For serotype 9V after the toddler dose the GMC ratio (13vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 1.13, 95% CI [0.95 to 1.33]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC After Toddler Dose vs 7vPnC/7vPnC After Toddler Dose; For serotype 14 after the toddler dose the GMC ratio (13vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/7vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 0.88, 95% CI [0.73 to 1.06]
Statistical Analysis 11: Comparison: 7vPnC/7vPnC After Toddler Dose vs 7vPnC/13vPnC After Toddler Dose; For serotype 14 after the toddler dose the GMC ratio (7vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/7vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 0.72, 95% CI [0.58 to 0.90]
Statistical Analysis 12: Comparison: 13vPnC/13vPnC After Toddler Dose vs 7vPnC/13vPnC After Toddler Dose; For serotype 14 after the toddler dose the GMC ratio (13vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 1.22, 95% CI [1.00 to 1.49]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC After Toddler Dose vs 7vPnC/7vPnC After Toddler Dose; For serotype 18C after the toddler dose the GMC ratio (13vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/7vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 0.82, 95% CI [0.69 to 0.97]
Statistical Analysis 14: Comparison: 7vPnC/7vPnC After Toddler Dose vs 7vPnC/13vPnC After Toddler Dose; For serotype 18C after the toddler dose the GMC ratio (7vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/7vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 0.86, 95% CI [0.69 to 1.08]
Statistical Analysis 15: Comparison: 13vPnC/13vPnC After Toddler Dose vs 7vPnC/13vPnC After Toddler Dose; For serotype 18C after the toddler dose the GMC ratio (13vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 0.95, 95% CI [0.78 to 1.15]
Statistical Analysis 16: Comparison: 13vPnC/13vPnC After Toddler Dose vs 7vPnC/7vPnC After Toddler Dose; For serotype 19F after the toddler dose the GMC ratio (13vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/7vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 1.26, 95% CI [1.00 to 1.59]
Statistical Analysis 17: Comparison: 7vPnC/7vPnC After Toddler Dose vs 7vPnC/13vPnC After Toddler Dose; For serotype 19F after the toddler dose the GMC ratio (7vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/7vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 0.91, 95% CI [0.68 to 1.20]
Statistical Analysis 18: Comparison: 13vPnC/13vPnC After Toddler Dose vs 7vPnC/13vPnC After Toddler Dose; For serotype 19F after the toddler dose the GMC ratio (13vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 1.39, 95% CI [1.08 to 1.79]
Statistical Analysis 19: Comparison: 13vPnC/13vPnC After Toddler Dose vs 7vPnC/7vPnC After Toddler Dose; For serotype 23F after the toddler dose the GMC ratio (13vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/7vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 0.81, 95% CI [0.67 to 1.00]
Statistical Analysis 20: Comparison: 7vPnC/7vPnC After Toddler Dose vs 7vPnC/13vPnC After Toddler Dose; For serotype 23F after the toddler dose the GMC ratio (7vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/7vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 0.85, 95% CI [0.67 to 1.07]
Statistical Analysis 21: Comparison: 13vPnC/13vPnC After Toddler Dose vs 7vPnC/13vPnC After Toddler Dose; For serotype 23F after the toddler dose the GMC ratio (13vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose / 7vPnC Infant Series/13vPnC Toddler Dose After Toddler Dose) was calculated; Test type: Superiority or Other; Ratio = 0.96, 95% CI [0.78 to 1.19]

4. Secondary Outcome: Percentage of Participants Achieving Antibody Titer ≥1:8 After the Toddler Dose in 13vPnC/13vPnC and 7vPnC/13vPnC Groups
Description: Percentage of participants achieving functional antibody titer ≥1:8 as measured by opsonophagocytic activity assay (OPA) along with the corresponding 95% CI for the 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after the toddler dose (at 13 months of age)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- 13vPnC/13vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with a vaccine containing Pentavac at 2, 3, and 4 months of age (infant series) and 12 months of age (toddler dose).
- 7vPnC/13vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with Pentavac at 2, 3, and 4 months of age (infant series). Participants received one single 0.5 mL dose of 13vPnC coadministered with Pentavac at 12 months of age (toddler dose).
Arm/Group | 13vPnC/13vPnC After Toddler Dose | 7vPnC/13vPnC After Toddler Dose
Number analyzed (Participants) | 241 | 121
Percentage of Participants
  Additional Serotypes - Serotype 1 | 100.0 [95.9 to 100.0] | 98.9 [94.0 to 100.0]
  Additional Serotypes - Serotype 3 | 100.0 [95.9 to 100.0] | 97.8 [92.2 to 99.7]
  Additional Serotypes - Serotype 5 | 100.0 [95.9 to 100.0] | 97.8 [92.2 to 99.7]
  Additional Serotypes - Serotype 6A | 100.0 [95.8 to 100.0] | 98.9 [94.0 to 100.0]
  Additional Serotypes - Serotype 7F | 100.0 [95.8 to 100.0] | 100.0 [95.9 to 100.0]
  Additional Serotypes - Serotype 19A | 98.8 [93.7 to 100.0] | 97.8 [92.2 to 99.7]

5. Secondary Outcome: Geometric Mean Titer (GMT) in 13vPnC/13vPnC and 7vPnC/13vPnC Groups After the Toddler Dose
Description: GMT as measured by opsonophagocytic activity assay (OPA) for 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after the toddler dose (at 13 months of age)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- 13vPnC/13vPnC After Toddler Dose: Subjects received one single 0.5 mL dose of 13vPnC coadministered with Pentavac at 2, 3, 4, and 12 months of age.
- 7vPnC/13vPnC After Toddler Dose: Subjects received one single 0.5 mL dose of 7vPnC coadministered with Pentavac at 2, 3, and 4 months. One single 0.5 mL dose of 13vPnC was coadministered with Pentavac at 12 months of age.
Arm/Group | 13vPnC/13vPnC After Toddler Dose | 7vPnC/13vPnC After Toddler Dose
Number analyzed (Participants) | 241 | 121
titer
  Additional Serotypes - Serotype 1 | 126.00 [99.87 to 158.97] | 61.58 [47.72 to 79.47]
  Additional Serotypes - Serotype 3 | 345.33 [296.06 to 402.80] | 428.88 [346.69 to 530.56]
  Additional Serotypes - Serotype 5 | 244.18 [200.14 to 297.92] | 130.99 [103.68 to 165.50]
  Additional Serotypes - Serotype 6A | 1346.83 [1143.98 to 1585.65] | 891.44 [694.76 to 1143.81]
  Additional Serotypes - Serotype 7F | 8126.24 [6657.36 to 9919.21] | 17034.59 [14316.59 to 20268.60]
  Additional Serotypes - Serotype 19A | 804.06 [615.90 to 1049.71] | 1072.43 [799.06 to 1439.32]

6. Primary Outcome: Geometric Mean Concentration (GMC) as Measured by Enzyme-linked Immunosorbent Assay (ELISA) for Diphtheria Toxoid and Tetanus Toxoid in 13vPnC Group Relative to 7vPnC Group
Time Frame: One month after the 3-Dose Infant Series (at 5 months of age) and the Toddler Dose (at 13 months of age)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Groups:
- 13vPnC After the Infant Series: Participants received one single 0.5 mL dose of 13vPnC coadministered with a vaccine containing Pentavac at 2, 3, and 4 months of age (infant series).
- 7vPnC After the Infant Series: Participants received one single 0.5 mL dose of 7vPnC coadministered with a vaccine containing Pentavac at 2, 3, and 4 months of age (infant series).
- 13vPnC After the Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with a vaccine containing Pentavac at 12 months of age (toddler dose).
- 7vPnC After the Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with a vaccine containing Pentavac at 12 months of age (toddler dose).
Arm/Group | 13vPnC After the Infant Series | 7vPnC After the Infant Series | 13vPnC After the Toddler Dose | 7vPnC After the Toddler Dose
Number analyzed (Participants) | 266 | 263 | 241 | 133
IU/mL
  Diphtheria | 0.19 [0.17 to 0.21] | 0.24 [0.22 to 0.27] | 2.09 [1.87 to 2.34] | 2.60 [2.26 to 2.99]
  Tetanus | 0.20 [0.18 to 0.22] | 0.21 [0.19 to 0.23] | 1.08 [0.94 to 1.24] | 1.25 [1.05 to 1.47]
Statistical Analysis 1: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Diphtheria the GMC ratio was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lower bound of the 2-sided, 95% CI for the GMC ratio (13vPnC group/7vPnC group) was >0.5 (2-fold criterion); Ratio = 0.77, 95% CI [0.66 to 0.90]
Statistical Analysis 2: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Tetanus the GMC ratio was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.94, 95% CI [0.82 to 1.08]
Statistical Analysis 3: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Diphtheria the GMC ratio was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.80, 95% CI [0.67 to 0.97]
Statistical Analysis 4: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Tetanus the GMC ratio was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.86, 95% CI [0.69 to 1.08]

7. Primary Outcome: Geometric Mean Concentration (GMC) for Haemophilus Influenzae Type b (Hib) in 13vPnC Group Relative to 7vPnC Group
Time Frame: One month after the 3-Dose Infant Series (at 5 months of age) and the Toddler Dose (at 13 months of age)
Population: Evaluable immunogenicity (per protocol) population adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations.
Measure: Number (95% Confidence Interval); unit: μg/mL
Arm/Group | 13vPnC After the Infant Series | 7vPnC After the Infant Series | 13vPnC After the Toddler Dose | 7vPnC After the Toddler Dose
Number analyzed (Participants) | 244 | 241 | 240 | 132
μg/mL | 1.28 [1.10 to 1.49] | 1.40 [1.19 to 1.64] | 12.15 [10.54 to 14.00] | 11.68 [9.66 to 14.13]
Statistical Analysis 1: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Hib (PRP) the GMC ratio was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.91, 95% CI [0.73 to 1.14]
Statistical Analysis 2: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Hib (PRP) the GMC ratio was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 1.04, 95% CI [0.82 to 1.32]

8. Primary Outcome: Geometric Mean Concentration (GMC) as Measured by Enzyme-linked Immunosorbent Assay (ELISA) for Poliomyelitis (Type 1, Type 2 and Type 3) in 13vPnC Group Relative to 7vPnC Group
Time Frame: One month after the 3-Dose Infant Series (at 5 months of age) and the Toddler Dose (at 13 months of age)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC After the Infant Series | 7vPnC After the Infant Series | 13vPnC After the Toddler Dose | 7vPnC After the Toddler Dose
Number analyzed (Participants) | 258 | 256 | 239 | 129
titer
  Polio Type 1 | 24.99 [21.37 to 29.23] | 28.33 [24.40 to 32.89] | 253.05 [207.15 to 309.11] | 250.56 [193.17 to 324.99]
  Polio Type 2 | 17.75 [15.07 to 20.92] | 21.55 [18.43 to 25.20] | 408.34 [338.94 to 491.95] | 415.20 [325.57 to 529.52]
  Polio Type 3 | 41.08 [34.08 to 49.52] | 52.95 [43.26 to 64.82] | 536.32 [436.46 to 659.02] | 638.18 [501.50 to 812.13]
Statistical Analysis 1: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Polio Type 1 the GMC ratio was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.88, 95% CI [0.71 to 1.09]
Statistical Analysis 2: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Polio Type 2 the GMC ratio was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.82, 95% CI [0.66 to 1.03]
Statistical Analysis 3: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Polio Type 3 the GMC ratio was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.78, 95% CI [0.59 to 1.02]
Statistical Analysis 4: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Polio Type 1 the GMC ratio was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 1.01, 95% CI [0.72 to 1.41]
Statistical Analysis 5: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Polio Type 2 the GMC ratio was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.98, 95% CI [0.72 to 1.34]
Statistical Analysis 6: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Polio Type 3 the GMC ratio was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.84, 95% CI [0.60 to 1.17]

9. Primary Outcome: Geometric Mean Concentration (GMC) as Measured by ELISA for Pertussis Toxin (PT) and Pertussis Filamentous Hemagglutinin (FHA) in 13vPnC Group Relative to 7vPnC Group
Time Frame: One month after the 3-Dose Infant Series (at 5 months of age) and the Toddler Dose (at 13 months of age)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: EU/mL
Arm/Group | 13vPnC After the Infant Series | 7vPnC After the Infant Series | 13vPnC After the Toddler Dose | 7vPnC After the Toddler Dose
Number analyzed (Participants) | 263 | 262 | 239 | 133
EU/mL
  Pertussis - FHA | 97.12 [89.84 to 104.98] | 111.23 [102.80 to 120.35] | 204.28 [185.65 to 224.79] | 241.08 [210.92 to 275.55]
  Pertussis - PT | 62.94 [58.80 to 67.38] | 68.20 [63.60 to 73.14] | 61.09 [56.19 to 66.40] | 61.70 [54.55 to 69.78]
Statistical Analysis 1: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Pertussis - FHA the GMC ratio was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.87, 95% CI [0.78 to 0.98]
Statistical Analysis 2: Comparison: 13vPnC After the Infant Series vs 7vPnC After the Infant Series; For Pertussis - PT the GMC ratio was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.92, 95% CI [0.84 to 1.02]
Statistical Analysis 3: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Pertussis - FHA the GMC ratio was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.85, 95% CI [0.72 to 1.00]
Statistical Analysis 4: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Pertussis - PT the GMC ratio was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.99, 95% CI [0.86 to 1.14]

10. Primary Outcome: Percentage of Participants Achieving a Pneumococcal Antibody Level ≥0.35µg/mL (ELISA) After the 3-Dose Infant Series of 13vPnC
Description: as for outcome 2
Time Frame: One month after the 3-Dose Infant Series (at 5 months of age)
Population: Evaluable immunogenicity (per protocol) population adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n) = number of participants with a determinate immunoglobulin G (IgG) antibody concentration to the given serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC: Participants received one single 0.5 mL dose of 13vPnC coadministered with a vaccine containing Pentavac at 2, 3, and 4 months of age (infant series).
Arm/Group | 13vPnC
Number analyzed (Participants) | 266
percentage of participants
  Common Serotypes - Serotype 4 (n=244) | 91.4 [87.1 to 94.6]
  Common Serotypes - Serotype 6B (n=241) | 72.6 [66.5 to 78.1]
  Common Serotypes - Serotype 9V (n=238) | 92.9 [88.8 to 95.8]
  Common Serotypes - Serotype 14 (n=236) | 94.9 [91.3 to 97.3]
  Common Serotypes - Serotype 18C (n=242) | 90.5 [86.1 to 93.9]
  Common Serotypes - Serotype 19F (n=241) | 97.9 [95.2 to 99.3]
  Common Serotypes - Serotype 23F (n=244) | 82.8 [77.5 to 87.3]
  Additional Serotypes - Serotype 1 (n=240) | 90.8 [86.5 to 94.2]
  Additional Serotypes - Serotype 3 (n=242) | 96.3 [93.1 to 98.3]
  Additional Serotypes - Serotype 5 (n=243) | 84.0 [78.7 to 88.3]
  Additional Serotypes - Serotype 6A (n=243) | 85.6 [80.5 to 89.8]
  Additional Serotypes - Serotype 7F (n=238) | 97.5 [94.6 to 99.1]
  Additional Serotypes - Serotype 19A (n=244) | 97.5 [94.7 to 99.1]

11. Primary Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions
Description: Local reactions were collected using an electronic diary. Tenderness (Tender)was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Swelling and redness were scaled as Any (swelling or redness present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (Sev) (>7.0 cm). Participants may be represented in more than 1 category.
Time Frame: During the 4-day period after each dose
Population: The safety population included all participants who received at least 1 dose of vaccine, (n) = number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: Percentage of Participants
Groups:
- 13vPnC Dose 1: Participants received one single 0.5 mL dose of 13vPnC coadministered with a vaccine containing Pentavac at 2 months of age (infant series).
- 7vPnC Dose 1: Participants received one single 0.5 mL dose of 7vPnC coadministered with a vaccine containing Pentavac at 2 months of age (infant series).
- 13vPnC Dose 2: Participants received one single 0.5 mL dose of 13vPnC coadministered with a vaccine containing Pentavac at 3 months of age (infant series).
- 7vPnC Dose 2: Participants received one single 0.5 mL dose of 7vPnC coadministered with a vaccine containing Pentavac at 3 months of age (infant series).
- 13vPnC Dose 3: Participants received one single 0.5 mL dose of 13vPnC coadministered with a vaccine containing Pentavac at 4 months of age (infant series).
- 7vPnC Dose 3: Participants received one single 0.5 mL dose of 7vPnC coadministered with a vaccine containing Pentavac at 4 months of age (infant series).
- 13vPnC/13vPnC Toddler Dose; 7vPnC/13vPnC Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with a vaccine containing Pentavac at 12 months of age (toddler dose).
- 7vPnC/7vPnC Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with a vaccine containing Pentavac at 12 months of age (toddler dose).
Arm/Group | 13vPnC Dose 1 | 7vPnC Dose 1 | 13vPnC Dose 2 | 7vPnC Dose 2 | 13vPnC Dose 3 | 7vPnC Dose 3 | 13vPnC/13vPnC Toddler Dose | 7vPnC/7vPnC Toddler Dose | 7vPnC/13vPnC Toddler Dose
Number analyzed (Participants) | 302 | 309 | 302 | 309 | 302 | 309 | 273 | 152 | 137
Percentage of Participants
  Tender-Any (n=256,257,223,225,210,206,189,96,89) | 38.3 | 38.5 | 33.2 | 42.2 | 36.2 | 32.0 | 50.3 | 44.8 | 64.0
  Tender-Sig (n=237,245,203,208,188,193,155,86,75) | 5.5 | 4.9 | 5.4 | 6.7 | 3.7 | 3.1 | 5.2 | 4.7 | 8.0
  Swelling-Any (n=254,256,226,235,217,219,185,99,97) | 41.3 | 38.7 | 50.0 | 54.5 | 48.4 | 51.1 | 53.5 | 57.6 | 59.8
  Swelling-Mild(n=249,255,223,232,213,214,181,99,95) | 36.9 | 35.7 | 46.6 | 51.3 | 44.6 | 45.8 | 48.1 | 55.6 | 57.9
  Swelling-Mod (n=243,246,207,208,193,194,159,88,82) | 14.4 | 9.3 | 14.0 | 14.4 | 14.0 | 16.0 | 19.5 | 15.9 | 20.7
  Swelling-Sev (n=235,244,199,203,184,188,152,87,73) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.7 | 0.0 | 0.0
  Redness-Any (n=256,260,236,241,226,223,187,106,99) | 44.5 | 46.9 | 53.4 | 58.1 | 55.8 | 59.2 | 66.8 | 60.4 | 63.6
  Redness-Mild(n=252,259,234,240,223,221,180,106,95) | 40.9 | 45.6 | 50.9 | 56.7 | 52.5 | 55.7 | 60.0 | 54.7 | 60.0
  Redness-Mod (n=241,245,205,206,190,192,165,87,79) | 9.5 | 3.7 | 7.3 | 6.8 | 8.9 | 12.5 | 24.2 | 18.4 | 20.3
  Redness-Sev (n=234,244,199,203,184,188,152,86,73) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.7 | 0.0 | 0.0

12. Primary Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events
Description: Systemic events (fever [fv] ≥ 37.5 degrees Celsius [C], fever ≥ 38 C but ≤ 39 C, fever >39 C but ≤ 40 C, fever > 40 C, decreased [decr] appetite, irritability, increased [incr] sleep, decreased sleep, hives, use of medication [med] to treat symptoms [sx], and use of medication to prevent symptoms) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: During the 4-day period after each dose
Population: The safety population included all subjects who received at least 1 dose of vaccine, (n) = number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: Percentage of Participants
Groups:
- 13vPnC Dose 2; 7vPnC Dose 2: Participants received one single 0.5 mL dose of 7vPnC coadministered with a vaccine containing Pentavac at 3 months of age (infant series).
- 7vPnC/13vPnC Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with Pentavac at 12 months of age (toddler dose).
Arm/Group | 13vPnC Dose 1 | 7vPnC Dose 1 | 13vPnC Dose 2 | 7vPnC Dose 2 | 13vPnC Dose 3 | 7vPnC Dose 3 | 13vPnC/13vPnC Toddler Dose | 7vPnC/7vPnC Toddler Dose | 7vPnC/13vPnC Toddler Dose
Number analyzed (Participants) | 302 | 309 | 302 | 309 | 302 | 309 | 273 | 152 | 137
Percentage of Participants
  Fv≥38°C,≤39°C(n=244,250,212,217,201,208,174,99,83) | 13.5 | 10.0 | 19.8 | 25.3 | 26.9 | 27.9 | 36.8 | 41.4 | 42.2
  Fv>39°C,≤40°C(n=238,245,201,205,184,191,153,89,73) | 0.8 | 0.4 | 1.0 | 2.4 | 0.5 | 1.6 | 4.6 | 2.2 | 4.1
  Fv >40°C (n=238,245,200,205,184,190,153,88,73) | 0.0 | 0.0 | 0.0 | 0.0 | 0.5 | 0.0 | 0.7 | 0.0 | 0.0
  Decr appetite(n=243,251,211,218,194,199,167,96,83) | 24.7 | 23.1 | 18.5 | 26.1 | 23.2 | 21.1 | 29.3 | 34.4 | 31.3
  Irritability (n=261,265,232,238,217,211,178,99,91) | 54.4 | 52.5 | 48.3 | 49.6 | 41.9 | 40.3 | 50.6 | 46.5 | 50.5
  Incr sleep (n=256,259,215,227,194,204,163,92,81) | 34.0 | 41.3 | 28.4 | 32.2 | 23.7 | 28.4 | 21.5 | 23.9 | 23.5
  Decr sleep (n=246,253,,215,218,203,196,168,93,81) | 28.0 | 20.6 | 26.5 | 27.1 | 25.1 | 20.9 | 26.2 | 22.6 | 30.9
  Med-treat sx(n=248,259,224,227,202,214,180,100,89) | 29.0 | 32.8 | 38.4 | 44.5 | 36.1 | 42.1 | 47.8 | 54.0 | 55.1
  Med-prevent sx(n=252,260,221,236,201,213,181,99,85 | 34.5 | 34.6 | 36.7 | 40.3 | 28.4 | 37.6 | 38.7 | 44.4 | 40.0

13. Primary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After the 3-Dose Infant Series of 13vPnC
Description: Antibody GMC for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMC (13vPnC) and corresponding 2-sided 95% confidence intervals (CI) were evaluated.
Time Frame: One month after the 3-Dose Infant Series (at 5 months of age)
Population: The evaluable immunogenicity (per protocol) population was the primary analysis population consisting of eligible subjects who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n) = number of participants with a determinate antibody concentration for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 13vPnC
Number analyzed (Participants) | 266
μg/mL
  Common Serotypes - Serotype 4 (n=244) | 1.29 [1.14 to 1.46]
  Common Serotypes - Serotype 6B (n=241) | 0.74 [0.62 to 0.89]
  Common Serotypes - Serotype 9V (n=238) | 1.15 [1.03 to 1.28]
  Common Serotypes - Serotype 14 (n=236) | 2.74 [2.38 to 3.16]
  Common Serotypes - Serotype 18C (n=242) | 1.42 [1.26 to 1.60]
  Common Serotypes - Serotype 19F (n=241) | 1.55 [1.42 to 1.70]
  Common Serotypes - Serotype 23F (n=244) | 0.92 [0.80 to 1.06]
  Additional Serotypes - Serotype 1 (n=240) | 1.21 [1.07 to 1.38]
  Additional Serotypes - Serotype 3 (n=242) | 1.25 [1.13 to 1.37]
  Additional Serotypes - Serotype 5 (n=243) | 0.93 [0.82 to 1.06]
  Additional Serotypes - Serotype 6A (n=243) | 0.94 [0.82 to 1.06]
  Additional Serotypes - Serotype 7F (n=238) | 1.93 [1.73 to 2.15]
  Additional Serotypes - Serotype 19A (n=244) | 2.10 [1.87 to 2.35]

ADVERSE EVENTS:
Groups:
- 13vPnC Infant Series: Participants received one single 0.5 mL dose of 13vPnC coadministered with a vaccine containing Pentavac at 2, 3, and 4 months of age (infant series). Adverse events were collected from dose 1 to approximately one month after dose 3.
- 7vPnC Infant Series: Participants received one single 0.5 mL dose of 7vPnC coadministered with a vaccine containing Pentavac at 2, 3, and 4 months of age (infant series). Adverse events were collected from dose 1 to approximately one month after dose 3.
- 13vPnC Post-Infant Series: Participants received one single 0.5 mL dose of 13vPnC coadministered with a vaccine containing Pentavac at 2, 3, and 4 months of age (infant series). Adverse events were collected from approximately one month after dose 3 to toddler dose.
- 7vPnC Post-Infant Series: Participants received one single 0.5 mL dose of 7vPnC coadministered with a vaccine containing Pentavac at 2, 3, and 4 months of age (infant series). Adverse events were collected from approximately one month after dose 3 to toddler dose.
- 13vPnC/13vPnC Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with a vaccine containing Pentavac at 12 months of age (toddler dose). Adverse events were collected for approximately one month after toddler dose.
- 7vPnC/7vPnC Toddler Dose; 7vPnC/ 13vPnC Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with a vaccine containing Pentavac at 12 months of age (toddler dose). Adverse events were collected for approximately one month after toddler dose.
- 13vPnC / 13vPnC 6-Month Follow-up: Participants received one single 0.5 mL dose of 13vPnC coadministered with Pentavac at 2, 3, and 4 months of age (infant series) and 12 months of age (toddler). Adverse events were collected for approximately six months after last visit.
- 7vPnC / 7vPnC 6-Month Follow-up: Participants received one single 0.5 mL dose of 7vPnC coadministered with Pentavac at 2, 3, and 4 months of age (infant series) and 12 months of age (toddler). Adverse events were collected for approximately six months after last visit.
- 7vPnC / 13vPnC 6-Month Follow-up: Participants received one single 0.5 mL dose of 7vPnC coadministered with Pentavac at 2, 3, and 4 months of age (infant series) and at 12 months of age (toddler). Adverse events were collected for approximately six months after last visit.
Arm/Group | 13vPnC Infant Series | 7vPnC Infant Series | 13vPnC Post-Infant Series | 7vPnC Post-Infant Series | 13vPnC/13vPnC Toddler Dose | 7vPnC/7vPnC Toddler Dose | 7vPnC/ 13vPnC Toddler Dose | 13vPnC / 13vPnC 6-Month Follow-up | 7vPnC / 7vPnC 6-Month Follow-up | 7vPnC / 13vPnC 6-Month Follow-up
Serious Adverse Events (participants affected / at risk) | 5/304 | 5/309 | 8/290 | 5/299 | 2/273 | 0/152 | 2/134 | 6/267 | 1/150 | 0/133
Other Adverse Events (participants affected / at risk) | 142/304 | 162/309 | 12/290 | 11/299 | 125/272 | 64/152 | 63/137 | 2/267 | 2/150 | 2/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC Infant Series (N=304) | 7vPnC Infant Series (N=309) | 13vPnC Post-Infant Series (N=290) | 7vPnC Post-Infant Series (N=299) | 13vPnC/13vPnC Toddler Dose (N=273) | 7vPnC/7vPnC Toddler Dose (N=152) | 7vPnC/ 13vPnC Toddler Dose (N=134) | 13vPnC / 13vPnC 6-Month Follow-up (N=267) | 7vPnC / 7vPnC 6-Month Follow-up (N=150) | 7vPnC / 13vPnC 6-Month Follow-up (N=133)
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC Infant Series (N=304) | 7vPnC Infant Series (N=309) | 13vPnC Post-Infant Series (N=290) | 7vPnC Post-Infant Series (N=299) | 13vPnC/13vPnC Toddler Dose (N=272) | 7vPnC/7vPnC Toddler Dose (N=152) | 7vPnC/ 13vPnC Toddler Dose (N=137) | 13vPnC / 13vPnC 6-Month Follow-up (N=267) | 7vPnC / 7vPnC 6-Month Follow-up (N=150) | 7vPnC / 13vPnC 6-Month Follow-up (N=133)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 6 | 13 | 0 | 0 | 3 | 1 | 3 | 0 | 0 | 0
Hypermetropia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 2 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infantile colic (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 17 | 16 | 0 | 0 | 3 | 3 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 10 | 13 | 0 | 1 | 5 | 7 | 4 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Milk allergy (Immune system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 25 | 39 | 0 | 2 | 8 | 3 | 2 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 23 | 32 | 0 | 0 | 5 | 4 | 9 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 8 | 19 | 2 | 0 | 10 | 5 | 4 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 14 | 5 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 6 | 12 | 2 | 0 | 8 | 6 | 4 | 0 | 0 | 0
Ear infection (Infections and infestations) | 5 | 8 | 1 | 0 | 16 | 6 | 5 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 3 | 9 | 0 | 0 | 7 | 0 | 2 | 0 | 0 | 0
Varicella (Infections and infestations) | 5 | 6 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 4 | 5 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinotracheitis (Infections and infestations) | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Roseola (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 2 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinolaryngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral skin infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dacryocystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema infectiosum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Genital candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Human herpesvirus 6 infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacteria stool identified (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Crying (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 3 | 1 | 1 | 1 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 13 | 8 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Child abuse (Social circumstances) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 98/256 | 99/257 | 0/0 | 0/0 | 95/189 | 43/96 | 57/89 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (any)=present at site of vaccination.
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 74/223 | 95/225 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (any)
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 76/210 | 66/206 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (any)
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 13/237 | 12/245 | 0/0 | 0/0 | 8/155 | 4/86 | 6/75 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (significant)=present and interfered with limb movement.
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 11/203 | 14/208 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (significant)
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 7/188 | 6/193 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (significant)
Induration (Any) (Skin and subcutaneous tissue disorders) | 105/254 | 99/256 | 0/0 | 0/0 | 99/185 | 57/99 | 58/97 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (any)=present at site of vaccination.
Induration (Any) (Skin and subcutaneous tissue disorders) | 113/226 | 128/235 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (any)
Induration (Any) (Skin and subcutaneous tissue disorders) | 105/217 | 112/219 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (any)
Induration (Mild) (Skin and subcutaneous tissue disorders) | 92/249 | 91/255 | 0/0 | 0/0 | 87/181 | 55/99 | 55/95 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (mild)=0.5 centimeters (cm) to 2.0 cm.
Induration (Mild) (Skin and subcutaneous tissue disorders) | 104/223 | 119/232 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (mild)
Induration (Mild) (Skin and subcutaneous tissue disorders) | 95/213 | 98/214 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (mild)
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 35/243 | 23/246 | 0/0 | 0/0 | 31/159 | 14/88 | 17/82 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (moderate)=2.5 cm to 7.0 cm.
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 29/207 | 30/208 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (moderate)
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 27/193 | 31/194 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (moderate)
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/235 | 0/244 | 0/0 | 0/0 | 1/152 | 0/87 | 0/73 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (severe) >7.0 cm.
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/199 | 0/203 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (severe)
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/184 | 0/188 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (severe)
Erythema (Any) (Skin and subcutaneous tissue disorders) | 114/256 | 122/260 | 0/0 | 0/0 | 125/187 | 64/106 | 63/99 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (any)=present at site of vaccination.
Erythema (Any) (Skin and subcutaneous tissue disorders) | 126/236 | 140/241 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (any)
Erythema (Any) (Skin and subcutaneous tissue disorders) | 126/226 | 132/223 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 — Infant Series Dose 3; Erythema (any)
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 103/252 | 118/259 | 0/0 | 0/0 | 108/180 | 58/106 | 57/95 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (mild)=0.5 cm to 2.0 cm.
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 119/234 | 136/240 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (mild)
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 117/223 | 123/221 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (mild)
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 23/241 | 9/245 | 0/0 | 0/0 | 40/165 | 16/87 | 16/79 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (moderate)=2.5 cm to 7.0 cm.
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 15/205 | 14/206 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (moderate)
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 17/190 | 24/192 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (moderate)
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/234 | 0/244 | 0/0 | 0/0 | 1/152 | 0/86 | 0/73 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (severe) >7.0 cm.
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/199 | 0/203 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (severe)
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/184 | 0/188 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (severe)
Fever ≥38°C but ≤39°C (General disorders) | 33/244 | 25/250 | 0/0 | 0/0 | 64/174 | 41/99 | 35/83 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever ≥38 degrees C but ≤39 degrees C
Fever ≥38°C but ≤39°C (General disorders) | 42/212 | 55/217 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever ≥38 degrees C but ≤39 degrees C
Fever ≥38°C but ≤39°C (General disorders) | 54/201 | 58/208 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever ≥38 degrees C but ≤39 degrees C
Fever >39°C but ≤40°C (General disorders) | 2/238 | 1/245 | 0/0 | 0/0 | 7/153 | 2/89 | 3/73 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >39 degrees C but ≤40 degrees C
Fever >39°C but ≤40°C (General disorders) | 2/201 | 5/205 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >39 degrees C but ≤40 degrees C
Fever >39°C but ≤40°C (General disorders) | 1/184 | 3/191 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever >39 degrees C but ≤40 degrees C
Fever >40°C (General disorders) | 0/238 | 0/245 | 0/0 | 0/0 | 1/153 | 0/88 | 0/73 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >40 degrees C
Fever >40°C (General disorders) | 0/200 | 0/205 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >40 degrees C
Fever >40°C (General disorders) | 1/184 | 0/190 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever >40 degrees C
Decreased appetite (General disorders) | 60/243 | 58/251 | 0/0 | 0/0 | 49/167 | 33/96 | 26/83 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased appetite
Decreased appetite (General disorders) | 39/211 | 57/218 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased appetite
Decreased appetite (General disorders) | 45/194 | 42/199 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased appetite
Irritability (General disorders) | 142/261 | 139/265 | 0/0 | 0/0 | 90/178 | 46/99 | 46/91 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Irritability
Irritability (General disorders) | 112/232 | 118/238 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Irritability
Irritability (General disorders) | 91/217 | 85/211 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Irritability
Increased sleep (General disorders) | 87/256 | 107/259 | 0/0 | 0/0 | 35/163 | 22/92 | 19/81 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Increased sleep
Increased sleep (General disorders) | 61/215 | 73/227 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Increased sleep
Increased sleep (General disorders) | 46/194 | 58/204 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Increased sleep
Decreased sleep (General disorders) | 69/246 | 52/253 | 0/0 | 0/0 | 44/168 | 21/93 | 25/81 | 0/0 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased sleep
Decreased sleep (General disorders) | 57/215 | 59/218 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased sleep
Decreased sleep (General disorders) | 51/203 | 41/196 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased sleep

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.